CLINICAL TRIAL: NCT00706914
Title: A Randomized, Double-Blind, Active-Controlled, Parallel-Group, Multicenter, 4-Week Pilot Study to Assess Symptoms in Stable, Moderate to Severe COPD Patients Taking Aclidinium Bromide 200 mcg Once Daily in Combination With Formoterol Fumarate Once or Twice Daily Versus Formoterol Fumarate Twice Daily
Brief Title: Comparison of Aclidinium Bromide and Formoterol Fumarate in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Actual sample size of 156 was sufficient to estimate the clinical outcomes.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAC-MD-24
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Pulmonary Disease; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease; COPD; COAD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Once-daily aclidinium/formoterol (Experimental): Aclidinium bromide 200 µg/ formoterol fumarate 12 µg fixed-dose combination (FDC) once-daily in the morning, plus placebo once-daily in the evening
  Interventions: Drug: Once-daily aclidinium/formoterol; Drug: Placebo to formoterol fumarate
- Morning aclidinium/formoterol plus evening formoterol (Experimental): Aclidinium bromide 200 µg/formoterol fumarate 12 µg FDC once-daily in the morning, plus formoterol fumarate 12µg once-daily in the evening
  Interventions: Drug: Once-daily aclidinium/formoterol; Drug: Once-daily formoterol fumarate
- Formoterol BID (Active Comparator): Formoterol fumarate 12 µg twice-daily (BID)
  Interventions: Drug: Twice-daily formoterol fumarate

INTERVENTIONS:
Drug: Once-daily aclidinium/formoterol — Inhaled aclidinium bromide 200 µg/formoterol fumarate 12 µg fixed-dose combination once-daily in the morning
  Arms: Morning aclidinium/formoterol plus evening formoterol; Once-daily aclidinium/formoterol
Drug: Twice-daily formoterol fumarate — Inhaled formoterol fumarate 12 µg twice-daily (BID)
  Arms: Formoterol BID
Drug: Placebo to formoterol fumarate — Inhaled placebo to formoterol fumarate once-daily in the evening
  Arms: Once-daily aclidinium/formoterol
Drug: Once-daily formoterol fumarate — Inhaled formoterol fumarate 12 μg once-daily in the evening
  Arms: Morning aclidinium/formoterol plus evening formoterol

SUMMARY:
This exploratory study will compare the efficacy of the fixed-dose combination (FDC) of aclidinium bromide and formoterol fumarate once daily in the morning and placebo once in the evening vs. the FDC once daily in the morning and formoterol fumarate once in the evening vs. formoterol fumarate twice daily. The study will assess pulmonary function and symptoms in patients with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe COPD
* Smoking history of greater or equal to 10 pack-years
* Diagnosis of stable moderate to severe COPD as defined by the GOLD Guidelines
* Postbronchodilator FEV1 from 30% to 79% of predicted values, inclusive
* Postbronchodilator FEV1/FVC ratio < 0.70

Exclusion Criteria:

* History or presence of asthma, allergic rhinitis, or exercise-induced bronchospasm
* Hospitalization for an acute COPD exacerbation in the 3 months prior to study entry
* Respiratory tract infection (including the upper respiratory tract) or COPD exacerbation in the 6 weeks prior to study entry
* Eosinophil count of at least 600 cells/mm3
* Long term oxygen therapy > 15 hours a day

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-06-30 (Actual); Primary Completion 2008-11-11 (Actual); Study Completion 2008-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (39):
- United States (39):
  - Forest Investigative Site, Tucson, Arizona
  - Forest Investigative Site, Fullerton, California
  - Forest Investigative Site, Lakewood, California
  - Forest Investigative Site, Rancho Mirage, California
  - Forest Investigative Site, Redlands, California
  - Forest Investigative Site, San Diego, California
  - Forest Investigative Site, San Jose, California
  - Forest Investigative Site, Stockton, California
  - Forest Investigative Site, Wheat Ridge, Colorado
  - Forest Investigative Site, Hartford, Connecticut
  - Forest Investigative Site, New Britain, Connecticut
  - Forest Investigative Site, Waterbury, Connecticut
  - Forest Investigative Site, DeLand, Florida
  - Forest Investigative Site, Panama City, Florida
  - Forest Investigative Site, Tamarac, Florida
  - Forest Investigative Site, Tampa, Florida
  - Forest Investigative Site, Atlanta, Georgia
  - Forest Investigative Site, Austell, Georgia
  - Forest Investigative Site, Blue Ridge, Georgia
  - Forest Investigative Site, Bowling Green, Kentucky
  - Forest Investigative Site, Hazard, Kentucky
  - Forest Investigative Site, North Dartmouth, Massachusetts
  - Forest Investigative Site, Rochester, Minnesota
  - Forest Investigative Site, Florissant, Missouri
  - Forest Investigative Site, Saint Charles, Missouri
  - Forest Investigative Site, St Louis, Missouri
  - Forest Investigative Site, Albany, New York
  - Forest Investigative Site, Charlotte, North Carolina
  - Forest Investigative Site, Cincinnati, Ohio
  - Forest Investigative Site, Columbus, Ohio
  - Forest Investigative Site, Medford, Oregon
  - Forest Investigative Site, Pittsburgh, Pennsylvania
  - Forest Investigative Site, East Providence, Rhode Island
  - Forest Investigative Site, Spartanburg, South Carolina
  - Forest Investigative Site, Dallas, Texas
  - Forest Investigative Site, McKinney, Texas
  - Forest Investigative Site, Midvale, Utah
  - Forest Investigative Site, Richmond, Virginia
  - Forest Investigative Site, Milwaukee, Wisconsin

REFERENCES:
- See also: lac-md-24-synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4065&filename=lac-md-24-synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 31 sites in the United States (US). All sites screened at least one patient and, of these 31 sites, three sites did not enroll any patients. The first patient was screened in March 2008 and the last patient visit was in February 2009.
Groups:
- Once-daily Aclidinium/Formoterol: Aclidinium bromide 200 μg and formoterol fumarate 12 μg fixed-dose combination once-daily in the morning plus placebo once every evening
- Morning Aclidinium/Formoterol Plus Evening Formoterol: Aclidinium bromide 200 μg and formoterol fumarate 12 μg fixed-dose combination once-daily in the morning plus formoterol fumarate alone 12 μg once every evening
- Formoterol BID: Formoterol fumarate 12 μg twice-daily (BID)
Period: Overall Study
Arm/Group | Once-daily Aclidinium/Formoterol | Morning Aclidinium/Formoterol Plus Evening Formoterol | Formoterol BID
Started | 63 | 62 | 31
Completed | 57 | 58 | 30
Not Completed | 6 | 4 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 0
Not completed — Protocol Violation | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Once-daily Aclidinium/Formoterol | Morning Aclidinium/Formoterol Plus Evening Formoterol | Formoterol BID | Total
Number analyzed (Participants) | 63 | 62 | 31 | 156
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (7.2) | 63.9 (9.0) | 62.2 (10.1) | 63.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 15 | 68
  Male | 35 | 37 | 16 | 88

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Average Nocturnal Symptom Scores
Description: Nocturnal Symptom Score Scale: 0 = None; 1 = Symptoms causing early awakening or awakening once during the night; 2 = Symptoms causing early awakening or awakening two or more times during the night; 3 = Symptoms causing awakening for most time during the night, 4 = Symptoms which were so severe that I could not sleep at all
Time Frame: Week 4 of treatment
Population: Includes the number of patients in the randomized population with available analysis value at both baseline and a specific time point. Randomized population defined as all patients in the screened population who were randomized to a treatment group in the study.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Once-daily Aclidinium/Formoterol | Morning Aclidinium/Formoterol Plus Evening Formoterol | Formoterol BID
Number analyzed (Participants) | 62 | 61 | 31
Units on a scale | -0.15 [-0.33 to 0.04] | -0.09 [-0.26 to 0.08] | -0.35 [-0.59 to -0.12]

2. Primary Outcome: Change From Baseline in Weekly Average Daily (24 Hour) Sputum Volume Scores
Description: Sputum Volume Score Scale: 0 = None; 1 = The amount of one teaspoon; 2 = The amount of one tablespoon; 3 = More than one tablespoon
Time Frame: Week 4 of treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Once-daily Aclidinium/Formoterol | Morning Aclidinium/Formoterol Plus Evening Formoterol | Formoterol BID
Number analyzed (Participants) | 62 | 61 | 31
Units on a scale | -0.17 [-0.34 to -0.01] | 0.13 [-0.07 to 0.32] | -0.00 [-0.20 to 0.20]

3. Other Pre Specified Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1)
Description: The trough value for each pulmonary function parameter was defined as the mean of the two greatest readings assessed 23 hours and 24 hours following the administration of the morning dose of the previous day
Time Frame: Week 4 of treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Once-daily Aclidinium/Formoterol | Morning Aclidinium/Formoterol Plus Evening Formoterol | Formoterol BID
Number analyzed (Participants) | 57 | 57 | 31
Liters | 0.097 [0.059 to 0.135] | 0.084 [0.040 to 0.128] | 0.118 [0.070 to 0.166]

4. Other Pre Specified Outcome: Change From Baseline in Peak Forced Expiratory Volume in One Second (FEV1)
Time Frame: Week 4 of treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Once-daily Aclidinium/Formoterol | Morning Aclidinium/Formoterol Plus Evening Formoterol | Formoterol BID
Number analyzed (Participants) | 62 | 61 | 31
Liters | 0.355 [0.308 to 0.403] | 0.319 [0.265 to 0.373] | 0.280 [0.220 to 0.341]

5. Other Pre Specified Outcome: Change From Baseline in Normalized Area Under the Curve (0-3 hr) of Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 values obtained at 30, 60, 120, and 180 minutes after the morning study drug dose
Time Frame: Week 4 of treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Once-daily Aclidinium/Formoterol | Morning Aclidinium/Formoterol Plus Evening Formoterol | Formoterol BID
Number analyzed (Participants) | 62 | 61 | 31
Liters | 0.257 [0.211 to 0.302] | 0.226 [0.176 to 0.276] | 0.200 [0.142 to 0.258]

ADVERSE EVENTS:
Time Frame: 29 ± 2 days
Arm/Group | Once-daily Aclidinium/Formoterol | Morning Aclidinium/Formoterol Plus Evening Formoterol | Formoterol BID
Serious Adverse Events (participants affected / at risk) | 1/63 | 1/62 | 0/31
Other Adverse Events (participants affected / at risk) | 0/63 | 0/62 | 2/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Once-daily Aclidinium/Formoterol (N=63) | Morning Aclidinium/Formoterol Plus Evening Formoterol (N=62) | Formoterol BID (N=31)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Drug withdrawal convulsions (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Once-daily Aclidinium/Formoterol (N=63) | Morning Aclidinium/Formoterol Plus Evening Formoterol (N=62) | Formoterol BID (N=31)
Nausea (Gastrointestinal disorders) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Due to early termination of the study, the actual sample size is different from the study design (200 patients)

Actual sample size was 156, but because this was an exploratory study, this was considered sufficient to estimate the clinical outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and sponsor.